CLINICAL TRIAL: NCT04183829
Title: Effects of Prior Induced Termination of Pregnancy on Complications and Pregnancy Outcomes.
Status: Recruiting | Type: Observational
Sponsor: National Research Institute for Family Planning, China (Other Government)
Responsible Party: Sponsor
Other Study IDs: No.2018-I2M-1-004
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Reproductive Health; Abortion
MeSH Terms: interventions — Abortion, Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: induced termination of pregnancy — Medically, induced termination of pregnancy (I-TOP) is defined as an intervention to voluntarily terminate a pregnancy (ie, induced abortion) by either surgical or medical means so it does not result in a live birth.

SUMMARY:
A prospective multicenter cohort study to evaluate effects of prior induced termination of pregnancy on complications and pregnancy outcomes.

DETAILED DESCRIPTION:
A prospective multicenter cohort study to evaluate effects of prior induced termination of pregnancy on complications and pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* women have induced abortion in early pregnancy (<12 weeks of gestation).
* permanent population and no tendency to move.
* normal language expression and understanding ability, able to understand research content.
* be able and willing to provide written informed consent and effective contact information, and be willing to cooperate with follow-up investigations.

Exclusion Criteria:

* above the age of 40
* with history of adverse pregnancy and childbirth

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: women who have induced abortion in early pregnancy (<12 weeks of gestation)
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
adverse pregnancy outcomes | 2028.6
  the rate of different adverse pregnancy outcomes

SECONDARY OUTCOMES:
Complications | 2020.6
  the rate of different complications

CONTACTS AND LOCATIONS:
Overall Officials: Pei Kaiyan, Principal Investigator — National Research Institute for Family Planning (NRIFP)
Locations (12):
- China (12):
  - Zhongshan Boai Hospital, Zhongshan, Guangdong
  - Zhangjiakou Maternal and Child Health Hospital, Zhangjiakou, Hebei
  - Daqing People's Hospital, Daqing, Heilongjiang
  - Changzhou Maternal and Child Health Hospital, Changzhou, Jiangsu
  - Yangzhou Maternal and Child Health Hospital, Yangzhou, Jiangsu
  - People's Hospital of Inner Mongolia Autonomous Region, Hohhot, Mongolia Autonomous
  - Qingdao Maternal and Child Health Hospital, Qingdao, Shandong
  - Zaozhuang Maternal and Child Health Hospital, Zaozhuang, Shandong
  - Taiyuan Maternal and Child Health Hospital, Taiyuan, Shanxi
  - Tanggu Maternal and Child Health Hospital, Tanggu, Tianjin Municipality
  - Chongqing Health Center for Women and Children, Chongqing
  - Shenzhen Luohu Maternity and Child Healthcare Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: Undecided